CLINICAL TRIAL: NCT05676723
Title: Assessment of the Determinants of the Thoracic Fluid Content Measured by the Bioimpedance-based Starling System in Critically Ill Patients
Brief Title: Thoracic Fluid Content by Bioimpedance-based Starling System
Acronym: TFC-Bio
Status: Completed | Type: Observational
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Professor, Bicetre Hospital
Other Study IDs: 2018-A02825-50
Record Dates: First submitted 2022-11-15; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Distress Syndrome; Hemodynamic Instability; Shock; Fluid Overload Pulmonary Edema
Keywords: Acute Respiratory Distress Syndrome; Shock; Hemodynamic Monitoring; Fluid Balance; Pulmonary Edema
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock; Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Starling system is a completely non-invasive hemodynamic monitoring technique. It is able to measure the thoracic fluid content (TFC). The TFC is supposed to reflect the total content of fluid in the thorax. Thus, TFC may include two of the variables that are commonly used for hemodynamic monitoring: the extravascular lung water (EVLW), and the global end-diastolic volume (GEDV). However, whether the TFC actually reflects GEDV and EVLW has not been clearly established. The objective of the study is to establish the determinants of TFC among hemodynamic variables including EVLW and GEDV.

DETAILED DESCRIPTION:
The Starling system is a completely non-invasive hemodynamic monitoring technique. It measures cardiac output through bioreactance. It also measures the mean transthoracic electric impedance (Z0) from which the thoracic fluid content (TFC) can be derived. The TFC is the only other variable that is provided by the system besides cardiac output and that is not inferred from it. The TFC is supposed to reflect the total content of fluid in the thorax and may include two of the variables that are commonly used for hemodynamic monitoring: the extravascular lung water (EVLW), which is the volume of lung edema, and the global end-diastolic volume (GEDV), which is a static index of cardiac preload. Cardiac preload is an important physiological variable; a prerequisite for TFC as a reflect cardiac preload would be that its changes are tightly linked to the changes in well-established markers of cardiac preload, as the GEDV measured by transpulmonary thermodilution, or the central venous pressure (CVP). Nevertheless, this has never been demonstrated. In addition, TFC includes the volume of EVLW, which is the volume of fluid contend in the lungs outside the pulmonary vessels. Nevertheless, the degree to which TFC is influenced by absolute values and changes in EVLW has never been established. The objective of the study is to establish the determinants of TFC among well-known hemodynamic variables including EVLW and GEDV, as well the value of TFC as a marker of cardiac preload and lung water.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y.o.
* Hospitalization in an ICU
* Monitoring by transpulmonary thermodilution already in place
* Decision by clinicians in charge to perform volume expansion by saline or fluid removal by diuretics infusion and/or ultrafiltration ("Fluid" group)
* Or presence of Acute Respiratory Distress Syndrome according to the Berlin definition ("ARDS" group)

Exclusion Criteria:

* Refusal to join the study
* In "Fluid" group, circulatory failure whose treatment cannot be postponed for ≥5 minutes (time required for the installation of Starling system).
* Impossibility to paste bioreactance electrodes properly in the skin of the thorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients, aged ≥ 18 y.o, monitored by transpulmonary thermodilution will enter the study if:
  * a decision by clinicians in charge to perform volume expansion by saline or fluid removal by diuretics infusion and/or ultrafiltration will be taken ("Fluid" group)
  * an Acute Respiratory Distress Syndrome (ARDS) will be diagnosed according to the Berlin definition ("ARDS" group)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
TFC as marker of cardiac preload or lung water | 6-9 months
  To investigate the relationship between TFC measured by bioimpedance and other variables offered by a system of hemodynamic monitoring based on TPTD (Transpulmonary Thermodilutions).

SECONDARY OUTCOMES:
Assessement of the determinants of the TFC measured by the Starling System | 6-9 months
  To establish the determinants of TFC among hemodynamic variables including EVLW and GEDV.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Kremlin-Bicetre, Le Kremlin-Bicêtre, Île-de-France Region, France